CLINICAL TRIAL: NCT03928080
Title: Self-detection and Professional Screening Strategies for Early Detection of Periodontitis: Diagnostic Accuracy of Bleeding on Brushing, Salivary Activated Matrix Metalloproteinase-8 (aMMP-8) and CDC/AAP Screening Questionnaire
Brief Title: Diagnostic Accuracy of Rapid Non-clinical Screening Tests for Early Detection of Periodontitis
Status: Completed | Type: Observational
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Clinical Professor, The University of Hong Kong
Other Study IDs: PhD20190130; HKUCTR-2631 (Registry Identifier: HKU Clinical Trial Registry)
Record Dates: First submitted 2019-04-14; First posted 2019-04-25 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Periodontitis; Gingivitis
Keywords: diagnostic accuracy; early detection; self-assessment; periodontitis
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva and mouth rinse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental cohort: Primary study to assess diagnostic accuracy
  Interventions: Diagnostic Test: Bleeding on brushing
- Confirmation cohort: Second cohort to confirm results from the first study on independent population
  Interventions: Diagnostic Test: Bleeding on brushing

INTERVENTIONS:
Diagnostic Test: Bleeding on brushing — Index tests are bleeding on brushing and aMMP-8 Gold standard: clinical diagnosis performed by specialist
  Other Names: aMMP-8

SUMMARY:
Gum disease is the 6th most prevalent disease of mankind. It is a non-communicable non-resolving inflammation; if untreated it leads to tooth loss and inability to chew properly. It is one of the top 80 human disease contributing 3.5 million years lived with disability and the major cause of increasing oral health costs. Addressing this major public health problem requires greater attention to prevention and early detection.

Gum disease cases in the population remain largely undetected because an affected individual does not feel the presence of gum disease and as a consequence people seek attention in the later stages of the disease once tooth loss has occurred.

In this study the investigators will compare different methods of screening for gum disease and compare them against a full professional examination. The investigators hope to be able to propose simple and effective methods for self-assessment that will allow people to suspect the presence of the disease before tooth loss occurs and thus allow early diagnosis and better treatment.

The whole study procedures consist 3 screening tests and the standard clinical examination. The screening tests involves:(1) a screening questionnaire; (2) a saliva test; (3) a toothbrushing test. Thereafter the participants will receive a standard clinical examination which is regarded as the gold standard for diagnosis of gum disease. Results of these tests will be compared with the standard clinical examination to assess the diagnostic accuracy of these tests.

The general aim of this program is to improve early detection of periodontitis in the population using a self-detection approach based on a toothbrush test as an early sign and a self-performed saliva test as a screening test for an individual to seek professional dental care early in the gum disease process.

The general hypothesis is that combining self-assessment of toothbrush test with a saliva test as an assessment of key inflammatory process underlying gum disease will increase the diagnostic accuracy of a screening approach in the population.

DETAILED DESCRIPTION:
Introduction:

Severe periodontitis is the 6th most prevalent disease of mankind. It is a non-communicable non-resolving inflammation and biofilm dysbiosis; if untreated it leads to tooth loss and masticatory dysfunction. It is: i) one of the top 80 human disease contributing 3.5 million years lived with disability, ii) a source of social inequality, iii) together with its major sequel - tooth loss - it is responsible for 88% of lost productivity from oral diseases (estimated at 54 billion USD), and iv) it is the major cause of escalating oral health costs ( 442 billion USD/year) that in advanced economies represent up to 10% of total medical expenses. Addressing this major public health problem requires greater attention to prevention and early detection.

Periodontitis cases in the population remain largely undetected due to lack of knowledge of early warning signs that can be self detected and to the fact that affected individuals adapt to life with increased degrees of disability as the disease progresses from an early stage (stage I) towards increasingly severe and invalidating stages (III-IV). Not unexpectedly, treatment outcomes improve with early detection while costs increase for later diagnosis due to the need for surgical intervention and rehabilitation of the teeth that have been lost. In partnership with the American Academy of Periodontology (AAP), the Centers for Disease Control and Prevention (CDC) in the United states, has validated a questionnaire (CDC/AAP questionnaire) for first step is important but its focus on more advanced disease, while appropriate to address individuals with more advanced disease, while appropriate to address individuals with more advanced disease towards specialist care, is unlikely to produce cost-effective health gains.

Spontaneous gingival bleeding or gingival bleeding upon tooth brushing (BoB) is a key sign of periodontitis with the potential to become a useful sentinel sign for self-detection. Surprisingly little is known about BoB and its relationship to professional assessment and diagnosis. Few studies have shown that it is highly sensitive to detect gingival inflammation but it has low to moderate specificity for periodontitis as it is shared by both gingivitis (superficial gum inflammation) and periodontitis. Its diagnostic performance, however, may be improved by combining it with salivary test able to discriminate between gingivitis and periodontitis. Salivary activated matrix metalloproteinase-8 (aMMP-8) is a biomarker associated with the inflammatory driven destruction of the periodontal ligament and alveolar characteristic of periodontitis; it has been shown to be able to discriminate between gingivitis and periodontitis in a point of care, professional setting.

The general aim of this program is to improve early detection of periodontitis in the population using a self-detection approach based on BoB as a sentinel sign and a consumer version of a point of care aMMP-8 test as a screening test for an individual to seek professional attention early in the periodontitis disease process.

Aims and Hypotheses to be Tested The aims of this diagnostic trial are to assess the diagnostic performance of: i) bleeding on brushing (BoB) as a sentinel sign, ii) salivary aMMP-8 as a biomarker, iii) a validated questionnaire alone and/or in combination for the early detection of periodontitis.

The general hypothesis is that combining self-assessment of a sentinel sign with a biomarker assessment of key inflammatory process underlying periodontitis will increase the diagnostic accuracy of a screening approach in the population.

Plan of Investigation (i) Subjects The study will involve two populations: i) a convenience sample of adult and elderly subjects reporting for oral health care at Prince Philip Dental Hospital and ii) a validation sample drawn from the Hong Kong adult and elderly population.

Study 1. Consecutive patients reporting to Prince Philip Dental Hospital reception clinic (screening and admission clinic) will be invited to participate.

Study 2. A validation sample will be drawn from a population of Hong Kong adult and elderly population in community and primary care settings. Subjects will be invited to participate and will be examined at the Clinical Research Center of the Prince Philip Dental Hospital.

The prevalence of different stages of periodontitis in the population is estimated at 8-12% for stage III-IV periodontitis and 28-32% for stage I-II periodontitis.

A sample size of 332 subjects has been estimated based on previous studies evaluating the area under the receiving operating curve (ROC curve) of the CDC/AAP questionnaire (0.68) and the ability to detect a 0.07 improvement with 80% power and p<0.05. A total of 400 subjects will be recruited in each trial to compensate for missing data.

(ii) Methods Consenting subjects will be subject to 3 sequential index tests in a specified sequence: i) they will be administered a validated Cantonese version of CDC/AAP questionnaire; ii) subjects will be instructed to perform a 30 second mouthwash with a standard buffer in order to collect a full mouth sample for aMMP-8 analysis. This will be quantitatively assessed with a point of care test. iii) Subjects will then be instructed to brush their teeth for 2 minutes and the obtained slurry (saliva) quantitatively analyzed for the presence of blood with a spectrophotometric test.

Positive CDC/AAP test will be defined based on the pattern of response to 5 questions according to the criteria specified by a previous study.

Positive BoB test will be defined by the subject's identification of traces of blood in the brushing slurry and later validated quantitatively with a spectrophotometric method based on hemoglobin concentrations.

Positive aMMP-8 test for periodontitis will be defined as a concentration of aMMP-8 > 20 ng/ml as determined with quantitative point of care lateral flow immunoassay.

After completion of the 3 experimental tests, subjects will undergo a full-mouth periodontal examination conducted by a trained and calibrated periodontal specialist who will determine the clinical diagnosis based on the 2017 international classification and case definition of periodontitis and gingivitis.

(iii) Study design Cross sectional diagnostic trial with independent blind comparison of experimental tests with a reference standard (professional diagnosis of periodontitis by a registered specialist in a clinical setting). First trial on a convenience sample of subjects reporting to Prince Philip Dental Hospital for oral health care, validation trial in a representative sample of the Hong Kong population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above.
* Having the ability to learn the standard toothbrushing method with artificial intelligence powered toothbrush.
* Ability and willingness to give written informed consent.

Exclusion Criteria:

* Edentulous mouth.
* Pregnant females.
* Having received professional periodontal treatment (other than supragingival cleaning) within the previous 12 months.
* Having received antibiotic medication within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a convenience sample of consecutive untreated subjects seeking dental care at Prince Philip Dental Hospital
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity measure | 1day
  Sensitivity of BoB, aMMP-8 and CDC/AAP screening questionnaires alone and in combination to correctly identify periodontitis cases at the time of completion of clinical examination
Specificity measure | 1day
  Specificity of BoB, aMMP-8 and CDC/AAP screening questionnaires alone and in combination to correctly identify periodontitis cases at the time of completion of clinical examination
The area under the receiver operating characteristic curve (AUC) measure | 1day
  The area under the receiver operating characteristic curve (AUC) of BoB, aMMP-8 and CDC/AAP screening questionnaires alone and in combination to correctly identify periodontitis cases at the time of completion of clinical examination
The post-test probability measure | 1day
  The post-test probability of BoB, aMMP-8 and CDC/AAP screening questionnaires alone and in combination to correctly identify periodontitis cases at the time of completion of clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD,PhD,MMSc, Principal Investigator — The University of Hong Kong
Locations (1):
- Prince Philip Dental Hospital, the Univerisity of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Blicher B, Joshipura K, Eke P. Validation of self-reported periodontal disease: a systematic review. J Dent Res. 2005 Oct;84(10):881-90. doi: 10.1177/154405910508401003. PMID 16183785
- [Result] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Result] Carra MC, Gueguen A, Thomas F, Pannier B, Caligiuri G, Steg PG, Zins M, Bouchard P. Self-report assessment of severe periodontitis: Periodontal screening score development. J Clin Periodontol. 2018 Jul;45(7):818-831. doi: 10.1111/jcpe.12899. Epub 2018 May 16. PMID 29611224
- [Result] Eke PI, Dye BA, Wei L, Slade GD, Thornton-Evans GO, Beck JD, Taylor GW, Borgnakke WS, Page RC, Genco RJ. Self-reported measures for surveillance of periodontitis. J Dent Res. 2013 Nov;92(11):1041-7. doi: 10.1177/0022034513505621. Epub 2013 Sep 24. PMID 24065636
- [Result] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Result] Izadi Borujeni S, Mayer M, Eickholz P. Activated matrix metalloproteinase-8 in saliva as diagnostic test for periodontal disease? A case-control study. Med Microbiol Immunol. 2015 Dec;204(6):665-72. doi: 10.1007/s00430-015-0413-2. Epub 2015 Apr 5. PMID 25841875
- [Result] Kallio P, Ainamo J, Dusadeepan A. Self-assessment of gingival bleeding. Int Dent J. 1990 Aug;40(4):231-6. PMID 2397955
- [Result] Kallio P. Self-assessed bleeding in monitoring gingival health among adolescents. Community Dent Oral Epidemiol. 1996 Apr;24(2):128-32. doi: 10.1111/j.1600-0528.1996.tb00829.x. PMID 8654034
- [Result] Leppilahti JM, Ahonen MM, Hernandez M, Munjal S, Netuschil L, Uitto VJ, Sorsa T, Mantyla P. Oral rinse MMP-8 point-of-care immuno test identifies patients with strong periodontal inflammatory burden. Oral Dis. 2011 Jan;17(1):115-22. doi: 10.1111/j.1601-0825.2010.01716.x. PMID 20659259
- [Result] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Result] Trombelli L, Farina R, Silva CO, Tatakis DN. Plaque-induced gingivitis: Case definition and diagnostic considerations. J Periodontol. 2018 Jun;89 Suppl 1:S46-S73. doi: 10.1002/JPER.17-0576. PMID 29926936
- [Derived] Bi M, Xie Y, Yu X, Li H, Pelekos G, Jin L, Li Y, Tonetti MS. Clinical Features Associated With Periodontal Case Misclassification by an Active Matrix Metalloproteinase-8 Point-of-Care Oral Rinse Test. J Clin Periodontol. 2025 Sep;52(9):1276-1287. doi: 10.1111/jcpe.14189. Epub 2025 Jun 3. PMID 40462486
- [Derived] Deng K, Zonta F, Yang H, Pelekos G, Tonetti MS. Development of a machine learning multiclass screening tool for periodontal health status based on non-clinical parameters and salivary biomarkers. J Clin Periodontol. 2024 Dec;51(12):1547-1560. doi: 10.1111/jcpe.13856. Epub 2023 Sep 11. PMID 37697491
- [Derived] Uy SNMR, Deng K, Fok CTC, Fok MR, Pelekos G, Tonetti MS. Food intake, masticatory function, tooth mobility, loss of posterior support, and diminished quality of life are associated with more advanced periodontitis stage diagnosis. J Clin Periodontol. 2022 Mar;49(3):240-250. doi: 10.1111/jcpe.13588. Epub 2022 Jan 20. PMID 34935175
- [Derived] Deng K, Pelekos G, Jin L, Tonetti MS. Gingival bleeding on brushing as a sentinel sign of gingival inflammation: A diagnostic accuracy trial for the discrimination of periodontal health and disease. J Clin Periodontol. 2021 Dec;48(12):1537-1548. doi: 10.1111/jcpe.13545. Epub 2021 Oct 4. PMID 34494292